CLINICAL TRIAL: NCT05471609
Title: Sustained Release Oral Formulation for Treatment of Parkinson's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Levodopa

STUDY DESIGN:
Intervention Model Description: 2 different assemblies with 2 different formulations (A, B) will be used.
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- levodopa/carbidopa oral formulation A (Experimental): LD/CD will be delivered using an oral device placed in the oral/buccal cavity (between cheek and gum of lower jaw) and delivers continuous release of CD and LD for both transmucosal and gastrointestinal absorption.
  Interventions: Drug: levodopa/carbidopa oral formulation A
- levodopa/carbidopa oral formulation B (Experimental): LD/CD will be delivered using an oral device placed in the oral/buccal cavity (between cheek and gum of lower jaw) and delivers continuous release of CD and LD for both transmucosal and gastrointestinal absorption.
  Interventions: Drug: levodopa/carbidopa oral formulation B

INTERVENTIONS:
Drug: levodopa/carbidopa oral formulation A — Outer sachet 100mg CD/100mg LD and inner sachet 0mg CD /300mg LD
  Arms: levodopa/carbidopa oral formulation A
Drug: levodopa/carbidopa oral formulation B — Outer sachet 100mg CD/0mg LD and inner sachet 0mg CD /400mg LD
  Arms: levodopa/carbidopa oral formulation B

SUMMARY:
Achieving sustained blood levels of carbidopa/levodopa has been a challenge in the treatment of PD and although levodopa remains the most commonly used drug, motor fluctuations remain a major disability especially in advanced Parkinson's disease. The aim of this study is to determine the efficacy of a novel oral carbidopa-levodopa formulation in achieving a sustained blood level of levodopa and carbidopa in normal volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy
* Are 18-65 years of age
* Are not currently taking medications regularly
* Able to fast 6 hours (water allowed)

Exclusion Criteria:

* Pregnancy
* Inability to fast

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-06-16 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Carbidopa/levodopa serum level Efficacy of the delivery method | 4 times, then every 60 mins for a total of 6 hours after administration (total of 9 blood samples)
  Carbidopa/levodopa serum level

CONTACTS AND LOCATIONS:
Overall Officials: Khalaf Bushara, MD,FRCP, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided